CLINICAL TRIAL: NCT03746821
Title: Biotin Urine Collection Study
Brief Title: Biotin Sample Collection Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PROTOCOL-1001
Record Dates: First submitted 2018-11-08; First posted 2018-11-20 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers; Biotin Excretion
MeSH Terms: interventions — Biotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biotin (Other): Volunteers to take biotin suppliment
  Interventions: Dietary Supplement: Biotin

INTERVENTIONS:
Dietary Supplement: Biotin — Biotin supplements (2) to be taken daily

SUMMARY:
This protocol has been designed for a collection of urine samples from volunteers who will be given high dose biotin supplements over a period of 5 days, in order to provide a research sample bank to examine for biotin excretion rates

DETAILED DESCRIPTION:
This is a sample collection study from a minimum of 10 volunteers who will be required to take a Biotin supplement daily for a period of 5 days.

Each volunteer will be asked to read the volunteer information sheet and if they wish to participate in the study, the study admission form will be completed and the volunteer will be asked to sign a consent form.

After informed consent each volunteer will be assigned a unique volunteer number for the duration of the trial to provide anonymity. The volunteer will be provided with a daily diary, urine collection material and a full set of volunteer instructions.

The daily diary will collect the following information;

* Date
* Whether or not supplement was taken and time taken
* sample collection times during the day

Volunteers will be requested to:

Day 1: Collect a urine sample from every void during the day. Days 2-6: Take biotin supplements with their evening meal and collect a urine sample from every void during the day Day 7: Collect a urine sample from every void during the day

All samples will be stored in the SPD Bio-bank until required for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Willing to take biotin supplements and collect urine samples
* Has regular menstrual periods
* SPD employee or partner of SPD employee

Exclusion Criteria:

* Taking any other supplements or medication (other than contraceptive pill)
* Taken Antibiotics in the last 4 weeks
* Diagnosed with metabolic disorder, kidney or liver disease
* Known Pregnancy or seeking to conceive
* Breast feeding
* Undergoing medical investigation for hormone imbalance
* Condition that contra-indicates pregnancy
* Condition that contra-indicates use of biotin supplements

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Biotin excretion | 2 months
  rate of biotin excretion in urine

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Dr, Study Director — SPD Development company Ltd.
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
sample collection study only